CLINICAL TRIAL: NCT01339793
Title: Exploring the Relationships Among Hospital's Corporate Social Responsibility, Job Attitudes and Job Performance
Status: Completed | Type: Observational
Sponsor: Taipei Medical University WanFang Hospital (Other)
Responsible Party: Huei-Yin Chou, Department of Health Business Administration, Meiho University
Other Study IDs: 99080
Record Dates: First submitted 2011-04-20; First posted 2011-04-21 (Estimated); Last update posted 2011-04-29 (Estimated); Status verified 2011-04

CONDITIONS: Corporate Social Responsibility(CSR)
Keywords: corporate social responsibility; social identity theory; stakeholder theory; organizational commitment; organizational performance

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
In recent years, many hospitals have progressively perceived the importance of corporate social responsibility (CSR). More and more hospital superintendents thus have realized that they should have a CSR strategy to deal with various stakeholders. Hospital, as a health care sector, is a labor-intensive industry. The management of hospitals should view its employees as salient stakeholders as well as a sort of precious asset by which hospital can possess a unique competition advantage in the operation. It is therefore important for superintendent to understand an employee's perspective on CSR and its impact on employees' work attitudes and organizational performance.

DETAILED DESCRIPTION:
Based on the stakeholder theory and social identity theory, this study attempts to employ a survey approach to understand the superintendents and employees' perceptions of CSR, and to explore the effects of CSR on organizational commitment of employees and organizational performance. The samples are taken from the senior managers (such as the superintendent and vice superintendent) and employees in the hospitals of which the number of beds are more than 200. The structural equation modeling (SEM) is applied to confirm the research framework and to test the hypotheses. The results will provide a reference for the management and regulators of hospitals to set up the CSR policies, and contribute to senior managers on the CSR strategy and human resource development with regard to hospitals.

ELIGIBILITY:
Inclusion Criteria:

* senior managers (such as the superintendent and vice superintendent) and employees in the hospitals

Exclusion Criteria:

* none

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: employees in the hospitals
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2011-01; Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Huei-Yin Chou, Principal Investigator — Meiho University
Locations (1):
- Meiho University, Neipu, Pingtung, Taiwan